CLINICAL TRIAL: NCT04817826
Title: TremelImumab aNd Durvalumab Combination For the Non-operatIve Management (NOM) of Microsatellite InstabiliTY (MSI)-High Resectable Gastric or Gastroesophageal Junction Cancer: The Multicentre, Single-arm, Multi-cohort, Phase II INFINITY Study.
Brief Title: TremelImumab aNd Durvalumab For the Non-operatIve Management (NOM) of MSI-high Resectable GC/GEJC.
Acronym: INFINITY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003440-92
Record Dates: First submitted 2021-03-11; First posted 2021-03-26 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; Microsatellite Instability
Keywords: Durvalumab; Tremelimumab; Non-operative management; Surgery; Gastric cancer; Microsatellite Instability
MeSH Terms: conditions — Stomach Neoplasms; Microsatellite Instability | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Phase II, multicentre, single-arm, multi-cohort trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Pre-operative treatment with tremelimumab 300 mg single administration (day 1) and durvalumab 1500 mg Q4W for 3 cycles (day 1, 29 and 57).
  Patients in Cohort 1 will undergo standard gastrectomy with D2 lymphadenectomy and then they will be followed by an active follow-up every 12 weeks for two years and then a standard follow-up every six months until the end of the fifth year from surgery.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Cohort 2 (Experimental): Pre-operative treatment with tremelimumab 300 mg single administration (day 1) and durvalumab 1500 mg Q4W for 3 cycles (day 1, 29 and 57).
  In Cohort 2, patients with no evidence of complete clinical response will undergo standard gastrectomy with D2 lymphadenectomy and then they will be followed up. Patients with complete clinical response will undergo a non-operative management (NOM) with an active follow-up phase every 12 weeks for two years, followed by standard follow-up every six months until the end of the fifth year. At any time during follow-up, in case of clinical suspicion or confirmation of residual gastric cancer, patients will undergo standard surgery according to the clinical practice at their Centre.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — durvalumab 1500 mg Q4W for 3 cycles (day 1, 29 and 57).
Drug: Tremelimumab — tremelimumab 300 mg single administration (day 1)

SUMMARY:
INFINITY is a Phase II, multicentre, single-arm, multi-cohort trial aimed at evaluating the activity and safety of the combination of tremelimumab and durvalumab as neoadjuvant (Cohort 1) and definitive (Cohort 2) treatment for MSI-high gastric/gastroesophageal juction cancer patients eligible for radical surgery.

DETAILED DESCRIPTION:
This study will pre-screen approximately 310 patients, in order to enrol a total number of 31 patients, 18 in Cohort 1 and 13 in Cohort 2, across 25 Italian Centres.

After central confirmation of MSI-high, dMMR and EBV-negative status, patients with resectable gastric or gastroesophageal junction cancer (Siewert II/III), categorized as cT≥2, any cN, M0 or any cT, cN1-3, M0 according to TNM classification 8th edition, will be enrolled and they will receive a pre-operative treatment with tremelimumab 300 mg single administration (day 1) and durvalumab 1500 mg Q4W for 3 cycles (day 1, 29 and 57).

All patients will undergo a complete disease restaging with chest-abdomen-pelvis CT scan, 18-FDG PET/CT, EUS with biopsies and liquid biopsy.

In Cohort 1, patients will undergo standard gastrectomy with D2 lymphadenectomy between weeks 15 and 18 from enrolment (at least six weeks after the last treatment administration), followed by an active follow-up every 12 weeks for two years and then a standard follow-up every six months until the end of the fifth year from surgery. In Cohort 2, patients with no evidence of complete clinical response (defined as absence of disease persistence at radiological imaging, liquid biopsy and EUS) will be treated as in Cohort 1. Patients with complete clinical response will undergo a non-operative management (NOM) and will start an active follow-up phase every 12 weeks for two years with chest-abdomen-pelvis CT with contrast, 18-FDG PET/TC, if clinically indicated by the Investigator, EUS with multiple random biopsies of the tumor site and FNA of clinically suspicious regional nodes and liquid biopsy, followed by standard follow-up every six months until the end of the fifth year. At any time during follow-up, in case of clinical suspicion or confirmation of residual gastric cancer, either at imaging, pathologically at tissue biopsies/cytological specimens or at ctDNA in liquid biopsy, the patients will undergo standard surgery according to the clinical practice at their Centre (subtotal/total gastrectomy with D2 lymphadenectomy).

Enrolment in Cohort 2 will start only after the completion of enrolment in Cohort 1 and after the extensive evaluation of the final results of Cohort 1 regarding to all endpoints (including exploratory endpoints) and after potential amendment(s) on study design, eligibility criteria and study procedures requested by the Sponsor's Steering Committee and an Independent Data Monitoring Committee made of foreign experts, and after the approval of the Ethics Committee and the Italian Medicines Agency.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally required authorization (such as the European Union [EU] Data Privacy Directive) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years old.
3. ECOG Performance Status 0-1.
4. Body weight >30 kg.
5. Diagnosis of resectable gastric or gastroesophageal junction (Siewert II-III) cancer, categorized according to TNM classification 8th edition:

   * cT ≥ 2, any cN, M0
   * Any cT, cN1-3, M0
6. Absence of distant metastases as defined by negativity of computed tomography (CT) and 18-fluorodeoxyglucose positron-emission tomography (18-FDG PET).
7. Life expectancy of at least 12 weeks
8. MSI-high status confirmed by IHC and multiplex PCR, and EBV-negative status by ISH, as determined centrally at the Co-ordinating Centre. Lack of heterogeneity of dMMR status as showed by lack of tumor cells showing concomitant expression of all 4 protein markers.
9. Adequate bone marrow and organ function, as defined by laboratory tests:

   1. Neutrophil count ≥ 1.5 x 10^3/μL
   2. Platelet count ≥ 100 x 10^6/μL
   3. Haemoglobin ≥ 9 g/dL
   4. Total bilirubin lower than 1.5 time the upper-normal limits (ULN) of the Institutional normal values
   5. AST (SGOT) and/or ALT (SGPT) < 2.5 x ULN
   6. Creatinine clearance (calculated according to Cockroft and Gault) > 40 mL/min or serum creatinine < 1.5 x ULN.
10. Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating Centre.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Participation in another clinical study with an investigational product during the last 12 months
4. Signs of distant metastases.
5. Prior medical treatments or irradiation for gastric cancer.
6. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
7. Previous treatments with immune checkpoint inhibitors targeting CTLA4, including tremelimumab, PD-1 or PD-L1, including durvalumab.
8. History of allergy or severe hypersensitivity reaction to monoclonal antibodies.
9. History of autoimmune diseases or history of organ transplantation that require immunosuppressive therapy. The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients with celiac disease controlled by diet alone
10. History of active primary immunodeficiency. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
11. Any condition requiring systemic treatment with corticosteroids at doses equal or superior to 10 mg daily of prednisone or equivalents, or other immunosuppressive drugs within 14 days from the inclusion in the study. The following medications are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
12. Administration of live vaccines within 4 weeks from the inclusion in the study. Note: Patients, if enrolled, should not receive live vaccine while receiving study drug(s) and up to 30 days after the last dose of study drug(s).
13. History of allogenic organ transplantation
14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
15. Women in pregnancy or lactation condition. Women with child-bearing potential or sexually-active men not willing to use adequate contraception during the whole study period.
16. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome of Cohort 1: Pathological complete response (ypT0N0) and negative ctDNA status | From the enrollment of the first patient in Cohort 1 up to 4 months from the enrollment of the last patient in Cohort 1
  Rate of patients (%) achieving both pathological complete response (ypT0N0) and negative ctDNA status after neoadjuvant immunotherapy in the intention-to-treat population of Cohort 1
Primary outcome of Cohort 2: 2-year complete response rate | From the enrollment of the first patient in Cohort 2 up to 2 years from the end of pre-operative treatment of the last patient enrolled in Cohort 2
  2-year complete response rate, defined as the absence of macroscopic or microscopic residual disease (locally, regionally and distantly) at radiological examinations, tissue and liquid biopsy, in absence of salvage gastrectomy.

SECONDARY OUTCOMES:
Patients' quality of life | For each Cohort, from the enrollment of the first patient up to 4 months from the last patient starting the pre-operative treatment phase
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EORTC QLQ-C30 For questions 1-28 of EORTC QLQ-C30 a 4-point scale is used. It scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. For the questions 29 and 30 of EORTC QLQ-C30 a 7-points scale is used. It scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Patients' quality of life | For each Cohort, from the enrollment of the first patient up to 4 months from the last patient starting the pre-operative treatment phase
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EORTC QLQ-STO22.
  For questions 31-52 of EORTC QLQ-STO22 a 4-point scale is used. It scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
Patients' quality of life | For each Cohort, from the enrollment of the first patient up to 4 months from the last patient starting the pre-operative treatment phase
  Quality of life will be assessed through Patient reported outcomes (PRO) instrument. EuroQol EQ-5D-5L.
  The EQ-5D-5L uses for first 5 questions qualitative multiple choice answers with NO SCALE. For the last questions, a score from 0 to 100 indicates from the worst to the best outcome.
3-year disease-free survival | For each Cohort, from the enrollment of the first patient up to 3 years from the enrollment of the last patient
  time from the enrollment in the study to the occurrence of disease relapse (local and/or distant), second gastric or gastroesophageal junction cancer primary, or death from any cause.
5-year overall survival | For each Cohort, from the enrollment of the first patient up to 5 years from the enrollment of the last patient
  time from the enrollment in the study to the occurrence of death.
Metastases-free survival | For each Cohort, from the enrollment of the first patient up to 5 years from the enrollment of the last patient
  time from the enrollment in the study to the first evidence of metastases or death from any cause.
Gastrectomy-free survival (Cohort 2 only) | From the enrollment of the first patient up to 5 years from the enrollment of the last patient
  time from the inclusion in the study to the occurrence of gastrectomy or death from any cause.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | For each Cohort, from the enrollment of the first patient up to 5 years from the enrollment of the last patient
  incidence of adverse events during the treatment and follow-up phases, assessed according to CTCAE v5.0.
Post gastrectomy complications | For each Cohort, from the enrollment of the first patient up to 1 year from the enrollment of the last patient
  Rate of post-gastrectomy complications following tremelimumab and durvalumab as pre-operative treatment strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pietrantonio, MD, Principal Investigator — Fondazione IRCCS - Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
The trial results concerning the primary, secondary and exploratory outcomes will be published according to the standard guidelines. IPD could eventually be requested to the Sponsor and Principal Investigator, who will carefully evaluate the formal and motivated request.

REFERENCES:
- [Background] Chalabi M, Fanchi LF, Dijkstra KK, Van den Berg JG, Aalbers AG, Sikorska K, Lopez-Yurda M, Grootscholten C, Beets GL, Snaebjornsson P, Maas M, Mertz M, Veninga V, Bounova G, Broeks A, Beets-Tan RG, de Wijkerslooth TR, van Lent AU, Marsman HA, Nuijten E, Kok NF, Kuiper M, Verbeek WH, Kok M, Van Leerdam ME, Schumacher TN, Voest EE, Haanen JB. Neoadjuvant immunotherapy leads to pathological responses in MMR-proficient and MMR-deficient early-stage colon cancers. Nat Med. 2020 Apr;26(4):566-576. doi: 10.1038/s41591-020-0805-8. Epub 2020 Apr 6. PMID 32251400